CLINICAL TRIAL: NCT01879800
Title: One-Day Acceptance and Commitment Training Intervention in Primary Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lilian N. Dindo (Other)
Responsible Party: Sponsor-Investigator, Lilian N. Dindo, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201207748
Record Dates: First submitted 2013-05-30; First posted 2013-06-18 (Estimated); Results first posted 2015-08-28 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Mood Disorders; Hypertension; Diabetes; Hypercholesterolemia
MeSH Terms: conditions — Mood Disorders; Hypertension; Diabetes Mellitus; Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Treatment As Usual/Waitlist (No Intervention): Treatment As Usual/Waitlist
- Acceptance and Commitment Therapy plus Illness Management (Experimental): Acceptance and Commitment Training plus Illness Management (ACT-IM) Patients in the ACT-IM group will attend a 1-day group workshop. Three broad areas will be covered: 1) Illness Management will cover the importance of physical and psychological self-care for the management of co-morbid depression/anxiety and vascular problems 2) Behavioral Change Training will involve i) teaching patients how to recognize ineffective patterns of behavior and habits, ii) exploring and setting life goals and those related to mental and physical health, and iii) promoting effective and committed actions to achieve these goals despite the urge to do otherwise; 3) Mindfulness and Acceptance Training will emphasize new ways of managing troubling thoughts, feelings, and physical sensations .
  Interventions: Behavioral: Acceptance and Commitment Therapy plus Illness Management

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy plus Illness Management
  Other Names: ACT-IM
  Arms: Acceptance and Commitment Therapy plus Illness Management

SUMMARY:
The goal of this study is to 1) examine the feasibility and acceptability of a one-day Acceptance and Commitment Training + Illness Management (ACT-IM) intervention in patients with comorbid vascular disease risk factors and depression or anxiety; and 2) to evaluate the effectiveness of this brief group intervention(ACT-IM), compared to Treatment-As-Usual (TAU) on the mental health and functioning of patients with co-morbid mood/anxiety and vascular disease risk factors. Patients with vascular disease risk factors will be identified by physicians in Family Practice or Internal Medicine, through chart review, or through advertisements. Those with vascular risk factors will be screened and assessed for symptoms of depression or anxiety. Patients who are experiencing significant depressive or anxiety symptoms and are interested in the treatment arm of the study will be randomized to the ACT-IM intervention or to TAU. Assessments of the following will take place both before and after the intervention: depression, anxiety, functioning, illness self-management, blood vessel health, and blood.

DETAILED DESCRIPTION:
There is no difference in the recruitment, consent, or enrollment process for the ACT-IM or the TAU group.

Patients with vascular disease risk factors will be identified by physicians in Family Practice or Internal Medicine, through chart review, or through advertisements. Those responding to advertisements or who have been referred by a physician will be invited to complete a screening phone call or to complete an on-line screening measure. Potentially eligible patients who were identified through chart review will first be sent a letter. This letter will be followed, at least one week later, by a phone call to assess for interest in the study and to provide information about the screening.

Participants who are eligible at screening will be contacted by the research team to discuss the study and answer any questions the patient may have. If the patient is interested in participating in the treatment arm of the study, an appointment will be scheduled for an in-person assessment.

At the in-person baseline assessment, participants will be provided with a detailed description of the study, consent will be obtained, and a 90-120 minute assessment will begin.

Initial Assessment:

* vitals(height, weight, blood pressure, temperature, pules, respiration rate.
* blood draw(to test blood fat, sugars, and inflammation (lipid panel (LIPP), glucose (GLU), hemoglobin A1C (A1C), and hsCRP). For this blood draw we ask that the participant not consume alcohol for 24 hours preceding the visit. We ask that this be a 12 hour fasting blood draw. We also ask that the participant not take their medications the day of the draw, prescription or otherwise. Once the blood draw is complete, they made take any medications they have.
* Noninvasive measure of blood vessel health (finger plethysmography) using EndoPAT**.
* Interview: Hamilton Rating Scale for Depression and Hamilton Rating Scale for Anxiety
* Self Report measures
* Medical charts only to confirm the diagnosis of vascular disease, hypertension, diabetes, or obesity from the chart.

At the end of the assessment, participants will be randomly assigned, using a 2:1 ratio, to either ACT-IM or TAU.

Treatment:

Patients in the ACT-IM group will attend a 1-day group workshop. Each ACT-IM group will be held at the University of Iowa Hospitals and Clinics, include 8-12 patients, and last 6 hours. The ACT-IM group will be conducted by 2 psychologists and the IM portion will be completed by a physician with expertise in vascular disease-psychiatric comorbidity. Three broad areas will be covered: 1) Illness Management will cover the importance of physical and psychological self-care for the management of co-morbid depression/anxiety and vascular problems (e.g. fatigue, stress, poor nutrition management, and inadequate physical activity); 2) Behavioral Change Training will involve i) teaching patients how to recognize ineffective patterns of behavior and habits, ii) exploring and setting life goals and those related to mental and physical health, and iii) promoting effective and committed actions to achieve these goals despite the urge to do otherwise; 3) Mindfulness and Acceptance Training will emphasize new ways of managing troubling thoughts, feelings, and physical sensations (e.g., learning how to recognize, and develop cognitive distance from unhelpful thoughts such as "I can't take this anymore" and learning how to willingly face experiences that cannot be changed). In-session exercises and practice will be heavily emphasized during the group intervention. A manual with information about topics covered during the group will be distributed for home use. Lunch will be provided and breaks will be offered to minimize fatigue.

Two to four weeks after the intervention, the ACT-IM participants will be contacted by one of the PI's and asked to provide qualitative feedback about the workshop.

Follow up assessments will take place at 2-, 6-, 12-, and 24-weeks. The 2-week and 6-week follow-ups can be completed by phone or web and take 45-60 minutes.

The 12-week follow-up will include interview assessments of depression and anxiety and will be completed over the phone.

The 24-week assessment will replicate the baseline visit. Thus, it will be an in-person visit, lasting 90-120 minutes.

All interviews and interventions will be audio taped for: 1) assessment of treatment integrity (i.e., to ensure that therapists are following study procedures) and 2) for inter-rater reliability of the interview measures.

**At baseline and 6 month follow-up, participants will undergo non-invasive testing of endothelial cell function using the Endothelial Peripheral Arterial Tone (EndoPAT). The EndoPAT is a medical device based on noninvasive Peripheral Arterial Tone (PAT)signal technology. It measures endothelium-mediated changes in vascular tone using unique bio-sensors placed on the fingertips. These changes in arterial tone are elicited by creating a down-stream hyperemic response induced by a standard 5-minute occlusion of the feeding artery (using a standard blood pressure cuff). When the cuff is released, the surge of blood flow causes an endothelium-dependent Flow-Mediated Dilation (FMD). The dilation or reactive hyperemia is captured by EndoPAT as an increase in the PAT Signal amplitude. A post-occlusion to pre-occlusion ratio is automatically calculated by the EndoPAT software, thus providing the EndoScore. Measurements from the opposite arm are used to control for concurrent non-endothelial dependent changes in vascular tone. Participants will be asked to clip their index fingernails before the visit or a research assistant may clip their fingernails before the study using sterilized clippers. Fingernails may need to be clipped if they are too long for the probes.

ELIGIBILITY:
Inclusion Criteria:

* The subject population is people ages 18-75 who have vascular risk factors (hypertension, diabetes mellitus or impaired fasting glucose, dyslipidemia, or obesity) and symptoms of depression or anxiety. Symptoms of depression and anxiety will be operationally defined as a score of >= 10 on the Patient Health Questionnaire (PHQ-8;depression) or GAD-7 (anxiety). All participants must be English speaking.

Exclusion Criteria:

* Patients with a primary psychotic disorder (e.g. schizophrenia).
* Patients with current alcohol or illicit drug dependence/abuse disorders.
* Patients who have started a new medication in previous 4 weeks or plan on starting a new medication in the next 4 weeks.
* Patients expressing active suicidal ideation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lilian N Dindo, PhD, Principal Investigator — University of Iowa; Jess Fiedorowicz, MD, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Acceptance and Commitment Therapy Plus Illness Management: Acceptance and Commitment Training plus Illness Management (ACT-IM) Patients in the ACT-IM group will attend a 1-day group workshop. Three broad areas will be covered: 1) Illness Management will cover the importance of physical and psychological self-care for the management of co-morbid depression/anxiety and vascular problems 2) Behavioral Change Training will involve i) teaching patients how to recognize ineffective patterns of behavior and habits, ii) exploring and setting life goals and those related to mental and physical health, and iii) promoting effective and committed actions to achieve these goals despite the urge to do otherwise; 3) Mindfulness and Acceptance Training will emphasize new ways of managing troubling thoughts, feelings, and physical sensations .
  Acceptance and Commitment Therapy plus Illness Management
Period: Overall Study
Arm/Group | Treatment As Usual/Waitlist | Acceptance and Commitment Therapy Plus Illness Management
Started | 14 | 30
Completed | 14 | 26
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment As Usual/Waitlist | Acceptance and Commitment Therapy Plus Illness Management | Total
Number analyzed (Participants) | 14 | 30 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 30 | 44
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: Years] | 45 [18 to 64] | 45 [18 to 64] | 45 [18 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 21 | 30
  Male | 5 | 9 | 14
Region of Enrollment [Number; unit: participants]
  United States | 14 | 30 | 44
Completed College [Number; unit: Participants]
  Completed College | 10 | 21 | 31
  Did Not Complete College | 4 | 9 | 13
Employed [Number; unit: Participants]
  Employed | 10 | 26 | 36
  Unemployed | 4 | 4 | 8
On Antidepressant medication [Number; unit: participants]
  On Antidepressants | 9 | 15 | 24
  Not on Antidepressants | 5 | 15 | 20

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Participants World Health Organization Quality of Life Measure- Physical Score: Change From Baseline to 3 and 6 Month Follow-up.
Description: The World Health Organization Quality of Life Measure- Physical scale assesses quality of life in physical health- specifically in activities of daily living, Dependence on medicinal substances and medical aids, Energy and fatigue, Mobility, Pain and discomfort, Sleep and rest, and Work Capacity. Outcome measure will be the change from baseline, at 3, and 6 months.
  Each item ranges in score from 1-5. Individual items are rated on a 5 point Likert scale where 1 indicates low, negative perceptions and 5 indicates high, positive perceptions. As such, domain and facet scores are scaled in a positive direction where higher scores denote higher quality of life.
  The mean score of the items within this physical domain is used to calculate the overall physical domain score. Mean scores are then multiplied by 4, yielding a score of 4 to 20. A higher domain score indicates a higher quality of life in physical ability.
Time Frame: Change at 3 and 6- Month Follow-up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Treatment As Usual/Waitlist | Acceptance and Commitment Therapy Plus Illness Management
Number analyzed (Participants) | 14 | 26
units on a scale
  3 Month Change from baseline | .85 (1) | 2.8 (.7)
  6 Month Change from baseline | 1.9 (1) | 4.1 (.7)

2. Secondary Outcome: Mean Change in Hamilton Depression Rating Scale (HAM-D) From Baseline to 3 and 6 Month Follow-up
Description: The HAM-D is a structured clinical interview for assessing depression severity. Outcome measure will be change from Baseline in Hamilton Depression Rating Scale and at 3 and 6 month follow-ups.
  Measure is scored by adding individual items and attaining an overall severity score. Scores range from 0 to 53, with higher values signifying a higher level of depression severity (and thus a worse outcome). A score of 0-7 is generally accepted to be within the normal range (or in clinical remission), while a score of 20 or higher (indicating at least moderate severity) is usually required for entry into a clinical trial.
Time Frame: 3-month and 6-Month Follow-Up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment As Usual/Waitlist | Acceptance and Commitment Therapy Plus Illness Management
Number analyzed (Participants) | 14 | 26
units on a scale
  3 month change from baseline | -2.8 (2.1) | -9.9 (1.4)
  6 month change from baseline | -.8 (2.5) | -11.7 (1.4)

3. Secondary Outcome: Mean Change in Hamilton Anxiety Rating Scale (HAM-A) From Baseline to 3 and 6 Month Follow-up
Description: The Hamilton Anxiety Rating Scale (HAM-A) is a psychological questionnaire used by clinicians to rate the severity of a patient's anxiety.
  Each item is scored independently based on a five-point, ratio scale. Upon the completion of the evaluation, the clinician compiles a total, composite score based upon the summation of each of the 14 individually rated items. This calculation will yield a comprehensive score in the range of 0 to 56. It has been predetermined that the results of the evaluation can be interpreted as follows. A score of 17 or less indicates mild anxiety severity. A score from 18 to 24 indicates mild to moderate anxiety severity. A score of 25 to 30 indicates a moderate to severe anxiety severity. Lastly, a score above 30 represents severe anxiety severity. The mean change in ratings will be assessed from baseline to 3 and 6 months follow up.
Time Frame: 3- and 6- Month Follow-Up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Treatment As Usual/Waitlist | Acceptance and Commitment Therapy Plus Illness Management
Number analyzed (Participants) | 14 | 26
units on a scale
  3 Month change from baseline | -2.8 (2.3) | -12.2 (1.6)
  6 month change from baseline | 0 (2.4) | -12.7 (1.6)

ADVERSE EVENTS:
Arm/Group | Treatment As Usual/Waitlist | Acceptance and Commitment Therapy Plus Illness Management
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/30
Other Adverse Events (participants affected / at risk) | 0/14 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No